CLINICAL TRIAL: NCT01193868
Title: Phase II/Pharmacodynamic Study of the γ-secretase Inhibitor RO4929097 in Patients Who Have Recently Completed Front-Line Chemotherapy for Advanced Non-small Cell Lung Cancer
Brief Title: RO4929097 in Treating Patients With Advanced Non-Small Cell Lung Cancer Who Have Recently Completed Treatment With Front-Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug production halted.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-01989; NCI-2010-01989 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000684242; MDA-2009-0649; 2009-0649 (Other: M D Anderson Cancer Center); 8506 (Other: CTEP); N01CM00039 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- RO4929097 (Experimental): Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Blood and tumor tissue samples are collected for pharmacogenetic, pharmacodynamic, and biomarker studies by IHC, FISH, and TUNEL assay.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well RO4929097 works in treating patients with advanced non-small cell lung cancer who have recently completed treatment with front-line chemotherapy. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess clinical activity of the gamma-secretase inhibitor RO4929097 in patients with non-small cell lung cancer (NSCLC) who have recently completed front-line chemotherapy for advanced disease.

II. To assess whether percent change in tumor size 6 weeks after initiation of RO4929097 correlates with tumor expression of Notch pathway markers and stem cell markers and/or with host genotype polymorphisms for selected components of the Notch pathway.

SECONDARY OBJECTIVES:

I. To assess whether response by RECIST criteria and TTF correlate with tumor expression of Notch pathway markers and stem cell markers and/or with host genotype polymorphisms for selected components of the Notch pathway.

II. To compare tumor expression of Notch pathway and stem cell markers in this patient population with expression of these markers in tumors from our tumor bank from chemo-naive NSCLC patient.

III. To correlate expression of Notch pathway markers with expression of stem cell markers.

IV. To correlate host genotype polymorphisms for selected components of the Notch pathway and other stem cell pathways with tumor expression of Notch pathway and stem cell markers.

V. To correlate the presence of tumor EGFR activating mutations with: a) notch expression, b) stem cell marker expression, and c) response to RO4929097.

VI. To assess change in expression of Notch pathway markers and stem cell markers over the 3 days of therapy in a subset of patients and to correlate this with: a) subsequent response to therapy and TTF, b) changes of each marker over the first 3 days of therapy with changes in the other markers of interest and with changes in level of tumor cell apoptosis by TUNEL assay.

VII. For patients in whom pre chemotherapy tissue can be obtained, we will compare the post chemotherapy (pre RO4929097) expression of Notch pathway and stem cell markers to those observed in the pre chemotherapy tissue.

OUTLINE:

Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood and tumor tissue samples are collected for pharmacogenetic, pharmacodynamic, and biomarker studies by IHC, FISH, and TUNEL assay.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer that is incurable (stage IV or malignant effusion or recurrent)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with CT scan with cuts at 2.5 or 5 mm
* Patients must have tumor amenable to core biopsy (or by incisional, excisional or punch biopsy) for research purposes; the collaborating interventional radiologists will make the determination whether or not the patient has a tumor amenable to biopsy and whether or not the patient is medically an appropriate candidate for tumor biopsy
* The patient must have received front line cytotoxic chemotherapy (combination or single agent, with or without the addition of targeted agents) for advanced NSCLC
* Patients will be eligible whether or not they have had a response or stable disease or progression of tumor on the front line cytotoxic therapy, and whether or not they have tumor progression in the interval between their front line therapy and initiation of therapy on this study
* Patients will also be eligible if they have received maintenance cytotoxic chemotherapy (eg pemetrexed) following completion of the front line chemotherapy, provided there had not been tumor progression between the end of the front line chemotherapy and the initiation of the maintenance chemotherapy
* Patients may also have received prior adjuvant chemotherapy or chemoradiotherapy with curative intent (followed by tumor recurrence or progression) before being given the front line therapy for advanced disease
* The last planned front-line therapy cycle or maintenance therapy cycle must have been administered >= 3 weeks (or >= 6 weeks after last therapy if it included a nitrosourea or mitomycin-C) and =< 8 weeks prior to initiation of therapy on this study, although they may be registered on study (prior to drug administration) any time from 0-8 weeks after last planned front-line chemotherapy (to permit correlative studies to be arranged before therapy starts)
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT) and ALT(SGPT) =< 3 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal
* Hemoglobin ≥ 9 g/dL
* Since all patients on this study will undergo tumor biopsy, the patient must have coagulation parameters in keeping with guidelines used by the Department of Interventional Radiology at MD Anderson Cancer Center to decide whether or not a patient is suitable for biopsy; specifically, the patient must have an INR =< 1.7 x upper limit of normal (ULN), and the patient must not have received aspirin or coumadin within the previous week or a therapeutic dose of a heparin product within the previous 24 hours
* The effects of RO4929097on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because Notch signal pathway inhibitors are known to be teratogenic, women of childbearing potential must use two forms of contraception (i.e., barrier contraception and one other method of contraception) from at least 4 weeks prior to initiation of therapy on this study, for the duration of study participation, and for at least 2 months post-treatment; while it is unknown how long after last drug administration drug that remains in the body would pose a risk to a subsequent pregnancy, the plasma half-life of the drug would suggest that it would probably only be for a few days; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 2 months after study participation, the patient should inform the treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); following initiation of therapy with RO4929097, a pregnancy test (serum or urine) will be administered every 3 weeks while on study; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator or designate must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097
* Patients with lung cancer may have false-positive pregnancy tests due to production of beta-HCG by tumor; patients with a positive pregnancy test who are unlikely to be pregnant may be considered for entry on this trial if they are deemed to be unlikely to be pregnant by an obstetrician or gynecologist and if the study sponsor is in agreement with their study entry
* Female patients of childbearing potential are defined as patients to whom any of the following apply:

  * Patients with regular menses
  * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had tubal ligation
* Female patients may be considered to NOT be of childbearing potential for the following reasons:

  * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
  * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
* Since there is a very small possibility that RO4929097 would reach high enough concentrations in semen of men participating in this study to pose a threat to a fetus being carried by their sexual partner, men participating in the study must also use 2 methods of contraception including 1 barrier method from the time of initiation of therapy on the study until 2 months after their last treatment on the study if their sexual partner has childbearing potential; if their sexual partner is already pregnant, 1 barrier method must be used to minimize the probability of exposure of the fetus to potentially toxic concentrations of RO4929097; while teratogenicity from exposure of a fetus to a drug in semen is a theoretical possibility, there has been little documentation of this for any agent in humans, and it has been documented in animals primarily only if the drug is present in semen at the time of fertilization; in addition, it is unknown how long the drug might remain detectable in semen; although the plasma half-life of the drug would suggest that its level in seminal fluids would probably be very low by a few days after last drug administration
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RO4929097, breastfeeding should be discontinued if the mother is treated with RO4929097
* With respect to patients with brain metastases, most drugs assessed reach concentrations in brain metastases or in primary brain tumors that are comparable to those in other tumor sites (although this has not yet been tested for RO4929097); furthermore, lung cancer brain metastases have response rates to systemic therapy that are comparable to response rates in metastases in other sites, after correcting for number of organ systems involved by tumor, survival is not substantially different for advanced NSCLC patients with vs without brain metastases, and risk of symptomatic CNS hemorrhage is not substantially higher in NSCLC patients with vs without brain metastases; brain metastases are very common in NSCLC; hence, patients with asymptomatic or minimally symptomatic brain metastases are eligible for this trial provided it is not anticipated that they will require any of the following over the course of their participation in the trial:

  * Corticosteroids for control of cerebral edema
  * Enzyme-inducing anticonvulsants
  * Radiotherapy, surgery or other local therapy for the brain metastases
* Patients must be able to swallow tablets

Exclusion Criteria:

* Patients may be registered on the protocol any time from 0-8 weeks after administration of last front-line therapy or maintenance therapy, but should not receive their first treatment on this study until 3-8 weeks after administration of last front-line therapy or maintenance therapy (or 6-8 weeks for prior nitrosoureas or mitomycin-C), and must have recovered adequately from adverse events to meet other eligibility criteria
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption
* Diarrhea > grade 1 despite appropriate therapy
* Patients who are serologically positive for hepatitis A, B or C are ineligible
* Patients with > grade 1 (by CTCAE criteria) hyponatremia or hypocalcemia (based on measurement of ionized calcium), despite appropriate medical management are excluded from this study, as are patients with hypophosphatemia (serum phosphate below the lower limit of normal for the institution), hypomagnesemia, (serum magnesium below the lower limit of normal), hypokalemia, or hyperkalemia (serum potassium outside normal limits) despite appropriate medical management
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy (with antibiotics, antiviral or antifungal agents), symptomatic congestive heart failure, unstable angina pectoris, angina at rest, a history of torsades des pointes, potentially life-threatening cardiac arrhythmias (patients are permitted to have chronic, stable atrial fibrillation, premature atrial or ventricular contractions, sinus tachycardia, provided the rate is controlled at < 115 per minute, and sinus bradycardia, provided the rate is > 50 per minute), myocardial infarction within the previous 3 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because RO4929097 is a Notch pathway inhibiting agent with the potential for teratogenic or abortifacient effects
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with RO4929097
* Cardiovascular: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Patients requiring drugs that are known to cause torsades des pointes and/or prolonged QTc intervals are excluded; patients requiring drugs with a possible but unproven association with torsades des pointes and/or QTc prolongation may be eligible, but will require additional electrocardiogram assessments
* Patients who have not recovered to < CTCAE grade 2 toxicities related to prior therapy are not eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Blumenschein, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 15, 2010 to June 29, 2012. Recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early as a result of discontinued production of the study drug.
Groups:
- RO4929097: Oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days
Period: Overall Study
Arm/Group | RO4929097
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RO4929097
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 65 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Response Rate by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Percentage of participants with response per RECIST version 1.1: Complete Response (CR):Disappearance all target lesions. Any pathological lymph nodes with reduction in short axis to <10 mm. Partial Response (PR): At least 30% decrease in sum of diameters of target lesions, reference baseline sum diameters. Progressive Disease (PD): At least 20% increase in sum of diameters of target lesions, reference smallest sum on study (includes baseline sum if that is smallest on study). In addition to relative increase of 20%, sum must demonstrate an absolute increase of at least 5 mm. (Note: appearance of 1 or more new lesions also considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum diameters while on study. Best response recorded from treatment start until disease progression/recurrence (reference for progressive disease the smallest measurements recorded since treatment started).
Time Frame: Response evaluation every 6 weeks (in addition to baseline scan, confirmatory scans approximately 6-7 (not less than 4) weeks following initial documentation of objective response). Expected follow up to 5 years, actual study period 9/2010 to 4/2014.
Population: Only those participants who have measurable disease present at baseline and received at least one dose of study medication considered evaluable for response with their response classified according to the RECIST definitions stated. Participants who exhibit objective disease progression prior to the end of cycle 1 also considered evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | RO4929097
Number analyzed (Participants) | 5
percentage of participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Progression (PD) | 100
  Stable Disease (SD) | 0

2. Primary Outcome: Percentage of Tumor Shrinkage as a Continuous Variable
Description: Response is reported as a continuous variable, as % change in tumor size from baseline. Pearson and Spearman correlation coefficients will be used. Reported with 95% two-sided confidence intervals.
Time Frame: 6 weeks
Population: Study terminated early with low accrual leading to insufficient data for analysis.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Tumors Expressing the Expression of Tumor Notch Markers and Stem Cell Markers of Interest in This Population vs Tumor Bank Population
Description: For participants having biopsies both before and after the agent, paired comparisons of post-therapy to pre-therapy results for the Notch IHC scores will be used. Researchers will assess changes from pre-therapy to post-therapy using a Wilcoxon Signed Rank Test (Wilcoxon rank sum tests). Spearman coefficients will be used to correlate tumor expression of Notch pathway markers with expression of stem cell markers.
Time Frame: Up to day 3
Population: Study terminated early with low accrual leading to insufficient data for analysis.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Tumors Expressing the Expression of Tumor Notch Markers and Stem Cell Markers of Interest in Participants With Versus Without a Particular Host Genotype Polymorphism
Description: Wilcoxon rank sum tests will be used. For participants having biopsies both before and after the agent, paired comparisons of post-therapy to pre-therapy results for the Notch IHC scores will be used. Researchers will assess changes from pre-therapy to post-therapy using a Wilcoxon Signed Rank Test (Wilcoxon rank sum tests).
Time Frame: Up to day 3
Population: Study terminated early with low accrual leading to insufficient data for analysis.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Tumors Expressing the Expression of Tumor Notch Markers and Stem Cell Markers of Interest in Participants With vs Without Epidermal Growth Factor Receptor (EGFR) Activating Mutations
Description: Wilcoxon rank sum tests will be used. Compared using Fisher Exact Tests. For participants having biopsies both before and after the agent, paired comparisons of post-therapy to pre-therapy results for the Notch IHC scores will be used. Researchers will assess changes from pre-therapy to post-therapy using a Wilcoxon Signed Rank Test (Sum Test). Spearman coefficients will be used to correlate tumor expression of Notch pathway markers with expression of stem cell markers.
Time Frame: Up to day 3
Population: Study terminated early with low accrual leading to insufficient data for analysis.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

6. Secondary Outcome: Proportion of Tumors Expressing the Expression of Tumor Notch Markers and Stem Cell Markers of Interest in Participants With vs Without Response by RECIST Criteria
Description: Wilcoxon rank sum tests will be used.
Time Frame: Up to day 3
Population: Study terminated early. Analysis not performed due to small numbers.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

7. Secondary Outcome: Proportion of Tumors Expressing the Expression of Tumor Notch Markers and Stem Cell Markers of Interest in Participants With vs Without Tumor Progression
Description: Tumor Immunohistochemistry (IHC) scores for Notch pathway and stem cell markers used in comparison to tumor progression; and progression evaluated in using international criteria proposed by revised RECIST guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. Wilcoxon rank sum tests will be used. Compared using Fisher Exact Tests.
Time Frame: Up to 3 months
Population: Study terminated early with low accrual leading to insufficient data for analysis.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

8. Secondary Outcome: Correlation of Tumor Shrinkage/Response With Biomarker Expression
Description: Correlate percent change in tumor size at 6 weeks (or at time off study, if therapy is stopped earlier due to tumor progression) with tumor Immunohistochemistry (IHC) scores for Notch pathway and stem cell markers; Tumor % shrinkage with RO4929097 will correlate with pre-therapy tumor expression of Notch pathway members, with expression of stem cell markers, and with changes in these over the first cycle of therapy.
Time Frame: 6 weeks
Population: Study terminated early. Analysis not performed due to small numbers.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

9. Secondary Outcome: Progression-free Survival
Description: Time from initiation of study drug until death, progression of tumor, or for worsening of tumor that did not meet RECIST 1.1 criteria but that did require discontinuation of therapy, assessed up to 5 years
Time Frame: Baseline up to 5 years
Population: Study terminated early. Analysis not performed due to small numbers.
Arm/Group | RO4929097
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events reporting includes events that occur within 30 days of the last dose of the investigational agent/treatment. Overall study period: 9/15/2010 to 6/20/2013.
Arm/Group | RO4929097
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO4929097 (N=6)
Death NOS (General disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO4929097 (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Blood bilirubin increased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5)
Hypotension (Vascular disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Pain (General disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study closed June 2012 with the NCI discontinuation production of the study drug RO4929097.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less